CLINICAL TRIAL: NCT00696514
Title: Vitamin B12 and Folic Acid Supplementation for Preventing Fractures in Elderly People
Acronym: B-PROOF
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Wageningen University (Other)
Collaborators: ZonMw: The Netherlands Organisation for Health Research and Development (Other); MCO Health (Unknown); Erasmus Medical Center (Other); Amsterdam UMC, location VUmc (Other); NZO: Dutch Dairy Association (Unknown)
Responsible Party: ZonMw: The Netherlands Organisation for Health Research and Development, ZonMw: The Netherlands Organisation for Health Research and Development
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: ZonMw 6130.0031; NTR1333
Record Dates: First submitted 2008-06-09; First posted 2008-06-12 (Estimated); Last update posted 2011-08-25 (Estimated); Status verified 2011-08

CONDITIONS: Osteoporosis; Cognitive Decline
Keywords: fracture; cognition
MeSH Terms: conditions — Osteoporosis; Cognitive Dysfunction; Fractures, Bone | interventions — Vitamin B 12; Folic Acid; Cholecalciferol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 2 (Placebo Comparator): placebo capsule, once per day
  Interventions: Dietary Supplement: Placebo (Vitamin D3) - 600 IU per day
- 1 (Experimental): Vitamin B12 and folic acid capsule, once a day
  Interventions: Dietary Supplement: Vitamin B12, folic acid, Vitamin D3

INTERVENTIONS:
Dietary Supplement: Vitamin B12, folic acid, Vitamin D3 — 500 µg vitamin B12; 0.4 mg folic acid; 600 IU vitamin D3 in one capsule, once per day
  Arms: 1
Dietary Supplement: Placebo (Vitamin D3) - 600 IU per day — 600 IU vitamin D3 in one capsule, once per day
  Arms: 2

SUMMARY:
It is hypothesized that vitamin B12 and folic acid supplementation reduces the number of incident fractures. The proposed study, a randomized placebo-controlled intervention trial, compares daily supplementation with folic acid (400 mcg) and vitamin B12 (500 mcg) to a placebo for a period of two years or longer in 3000 men and women aged 70 years and older, with initial basal plasma total homocysteine (tHcy) levels >= 15 micromol/L. Fracture incidence and time to fracture will be assessed and used as the efficacy measure.

Metabolic studies in a sub sample of the population will be included aiming to contribute to an understanding of the biological mechanisms underlying the associations found between markers of B-vitamin status and bone quality.

DETAILED DESCRIPTION:
Rationale: There is growing evidence that an elevated homocysteine level is a risk factor for fracture incidence. The most common cause of homocysteine elevation is poor vitamin B12 and folate status. It is hypothesized that supplementation with 500 µg vitamin B12 and 400 µg folic acid will reduce fracture incidence in elderly people Main objective: to determine the efficacy of oral supplementation with vitamin B12 and folic acid in the prevention of fractures Study design: The trial is a randomized double-blind placebo-controlled trial, with two arms in parallel (placebo versus supplement). The intervention comprises a period of two years, and will be targeted to 3000 elderly subjects with elevated homocysteine levels. The study will be performed in institutions or residences for older persons around Wageningen, Rotterdam and Amsterdam.

Study population: 3000 elderly subjects (70 years and older) with elevated homocysteine levels Intervention (if applicable): One group receives daily a tablet with 500 µg vitamin B12 and 400 ug folic acid and the other group receives daily a placebo tablet. In both tablets 15 µg (600 IU) of vitamin D is included as well.

Main study parameters/endpoints: Fracture incidence is the primary outcome measure Time to fracture will be calculated. It is expected that in the intervention group 34% less fractures will occur than in the placebo group.

Nature and extent of the burden and risks associated with participation, benefit and group relatedness: First, participants need to be recruited. This will be done via information letters. Those who are interested have to complete a small questionnaire and then they will receive an information brochure. Upon continued interest in the intervention study, participants will be invited for a blood sampling. This blood sampling will take place (nearby or) at the location where the participants live. Immediately after the blood sampling a run-in period will start. Blood will be checked on homocysteine levels. Only participants with elevated levels of homocysteine will be included in the study. Two to four weeks after the run-in period the intervention study will be implemented. At the start of this intervention study several measurements will be performed and several questionnaires will be completed together with the participant at home. During the whole study participants need to take daily one tablet and they have to complete calenders to monitor fracture incidence. At the end of the study, blood sampling will be performed and several measurements and questionnaires will be repeated again at home.

ELIGIBILITY:
Inclusion Criteria:

* 65 years and older; based on entry date into study;
* Fasting plasma Hcy level >= 12 µmol/L and < 50 µmol/L;
* No current or recent (<4 months) use of supplements with very high doses of B-vitamins;
* Competent to make own decisions;
* Persons with skin cancer are allowed to participate.
* Compliance to tablet intake > 85%

Exclusion Criteria:

* Participation in other intervention trials;
* Serious medical conditions, e.g. cancer diagnosis within the last 5 years or recent myocardial infarction;
* Immobilization (bedridden, wheelchair bound);

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 3000 (Estimated)
Dates: Start 2008-09; Primary Completion 2013-03 (Estimated); Study Completion 2013-03 (Estimated)

PRIMARY OUTCOMES:
Fractures | two years

SECONDARY OUTCOMES:
Cognitive decline | two years
Bone health | two years
Physical performance | two years
Quality of life | two years
Nutritional status | two years

CONTACTS AND LOCATIONS:
Overall Officials: Lisette CPGM de Groot, Prof, Principal Investigator — Wageningen University
Locations (3):
- Netherlands (3):
  - VU University Amsterdam, Institute for Health Sciences, Amsterdam
  - Erasmus MC, Rotterdam
  - Wageningen University, Wageningen

REFERENCES:
- [Derived] van Soest APM, van de Rest O, Witkamp RF, van der Velde N, de Groot LCPGM. The association between adherence to a plant-based diet and cognitive ageing. Eur J Nutr. 2023 Aug;62(5):2053-2062. doi: 10.1007/s00394-023-03130-y. Epub 2023 Mar 11. PMID 36905458
- [Derived] van Soest APM, van de Rest O, Witkamp RF, Cederholm T, de Groot LCPGM. DHA status influences effects of B-vitamin supplementation on cognitive ageing: a post-hoc analysis of the B-proof trial. Eur J Nutr. 2022 Oct;61(7):3731-3739. doi: 10.1007/s00394-022-02924-w. Epub 2022 Jun 15. PMID 35704085
- [Derived] Oliai Araghi S, Kiefte-de Jong JC, van Dijk SC, Swart KMA, van Laarhoven HW, van Schoor NM, de Groot LCPGM, Lemmens V, Stricker BH, Uitterlinden AG, van der Velde N. Folic Acid and Vitamin B12 Supplementation and the Risk of Cancer: Long-term Follow-up of the B Vitamins for the Prevention of Osteoporotic Fractures (B-PROOF) Trial. Cancer Epidemiol Biomarkers Prev. 2019 Feb;28(2):275-282. doi: 10.1158/1055-9965.EPI-17-1198. Epub 2018 Oct 19. PMID 30341095
- [Derived] van Dijk SC, Enneman AW, Swart KM, van Wijngaarden JP, Ham AC, de Jonge R, Blom HJ, Feskens EJ, Geleijnse JM, van Schoor NM, Dhonukshe-Rutten RA, de Jongh RT, Lips P, de Groot LC, Uitterlinden AG, van den Meiracker TH, Mattace-Raso FU, van der Velde N, Smulders YM. Effect of vitamin B12 and folic acid supplementation on biomarkers of endothelial function and inflammation among elderly individuals with hyperhomocysteinemia. Vasc Med. 2016 Apr;21(2):91-8. doi: 10.1177/1358863X15622281. Epub 2016 Jan 15. PMID 26774115
- [Derived] Brouwer-Brolsma EM, van der Zwaluw NL, van Wijngaarden JP, Dhonukshe-Rutten RA, in 't Veld PH, Feskens EJ, Smeets PA, Kessels RP, van de Rest O, de Groot LC. Higher Serum 25-Hydroxyvitamin D and Lower Plasma Glucose Are Associated with Larger Gray Matter Volume but Not with White Matter or Total Brain Volume in Dutch Community-Dwelling Older Adults. J Nutr. 2015 Aug;145(8):1817-23. doi: 10.3945/jn.115.214197. Epub 2015 Jul 1. PMID 26136594
- [Derived] van Wijngaarden JP, Dhonukshe-Rutten RA, van Schoor NM, van der Velde N, Swart KM, Enneman AW, van Dijk SC, Brouwer-Brolsma EM, Zillikens MC, van Meurs JB, Brug J, Uitterlinden AG, Lips P, de Groot LC. Rationale and design of the B-PROOF study, a randomized controlled trial on the effect of supplemental intake of vitamin B12 and folic acid on fracture incidence. BMC Geriatr. 2011 Dec 2;11:80. doi: 10.1186/1471-2318-11-80. PMID 22136481